CLINICAL TRIAL: NCT01002443
Title: Effect of Helicobacter Pylori Eradication on Glandular Atrophy and Intestinal Metaplasia in Patients Undergoing Subtotal Gastrectomy for Gastric Cancer
Brief Title: Efficacy Study of Helicobacter Pylori Eradication in Patients Undergoing Subtotal Gastrectomy for Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Il Ju Choi, M.D., Ph.D., National Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCCCTS03-063
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Gastric Cancer
Keywords: Helicobacter pylori; glandular atrophy; intestinal metaplasia; subtotal gastrectomy; gastric cancer; Precancerous lesion of gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H. pylori eradication (Active Comparator)
  Interventions: Drug: Helicobacter pylori eradication
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Helicobacter pylori eradication — Omeprazole 20 mg or Rabeprazole 10 mg bid + clarithromycin 500 mg and amoxicillin 1,000 mg bid for 7 days
  Arms: H. pylori eradication
Drug: placebo — Omeprazole 20 mg or Rabeprazole 10 mg bid + two placebo (for antibiotics) for 7 days
  Arms: placebo

SUMMARY:
Helicobacter pylori (H. pylori) is associated with gastric cancer in epidemiological studies.Gastric atrophy and intestinal metaplasia caused by H. pylori are considered as precancerous lesions, but whether H. pylori eradication improves these lesions is controversial.The primary objective of this study is to evaluate whether Helicobacter pylori eradication improves glandular atrophy and intestinal metaplasia which are known to be precancerous condition in patients undergoing subtotal gastrectomy for gastric cancer.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a primary etiological agent leading to chronic gastritis and peptic ulcer. The organism is also associated with gastric cancer in epidemiological studies. However, detailed mechanism of carcinogenesis remains unknown. Histolopathological studies indicate that chronic H. pylori infection progresses over decades through stages of chronic gastritis, atrophy, intestinal metaplasia, dysplasia and cancer. Gastric atrophy and intestinal metaplasia are considered as precancerous lesions, but whether H. pylori eradication improves these lesions is controversial. And the issue has not been evaluated in gastric cancer patients. However, despite the lack of evidence proven by a well-designed study, current guidelines from Europe and Japan recommend H. pylori eradication treatment in patients who were treated for gastric cancer by surgically or endoscopically. Thus, it is important to evaluate whether H. pylori eradication can improve known precancerous lesion, i.e. glandular atrophy and intestinal metaplasia in gastric cancer patients. Such histological improvement may eventually reduce secondary gastric cancer development and provide evidence for current guidelines. Helicobacter pylori is a primary etiological agent leading to chronic gastritis and peptic ulcer. The organism is also associated with gastric cancer in epidemiological studies. However, detailed mechanism of carcinogenesis remains unknown. Histolopathological studies indicate that chronic H. pylori infection progresses over decades through stages of chronic gastritis, atrophy, intestinal metaplasia, dysplasia and cancer. Gastric atrophy and intestinal metaplasia are considered as precancerous lesions, but whether H. pylori eradication improves these lesions is controversial. And the issue has not been evaluated in gastric cancer patients. However, despite the lack of evidence proven by a well-designed study, current guidelines from Europe and Japan recommend H. pylori eradication treatment in patients who were treated for gastric cancer by surgically or endoscopically. Thus, it is important to evaluate whether H. pylori eradication can improve known precancerous lesion, i.e. glandular atrophy and intestinal metaplasia in gastric cancer patients. Such histological improvement may eventually reduce secondary gastric cancer development and provide evidence for current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* AGC or EGC confirmed by endoscopy
* Histologically confirmed adenocarcinoma of stomach
* Helicobacter pylori infection was confirmed by biopsy and CLO
* Pre op CT stage: IA, IB, II, IIIA according to UICC TNM classification system
* Pre op biopsy (body LC side) shows either intestinal metaplasia or glandular atrophy (at least grade 1)
* Tumor location is suitable for subtotal gastrectomy- i.e. at or distal to lower body
* Informed consent should be signed

Exclusion Criteria:

* Recurrent gastric cancer
* Previous serious side effect to antibiotics
* H. pylori eradication treatment history
* Other malignancy within the past 5 years
* Pregnant or nursing women
* Serious concurrent infection or nonmalignant disease such as liver cirrhosis, renal failure, cardiovascular diseases
* Psychiatric disorder that would preclude compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2003-07; Primary Completion 2006-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Histological grading improvement rate | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, M.D., Ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- Research Institute and Hospital, National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Cho SJ, Choi IJ, Kook MC, Yoon H, Park S, Kim CG, Lee JY, Lee JH, Ryu KW, Kim YW. Randomised clinical trial: the effects of Helicobacter pylori eradication on glandular atrophy and intestinal metaplasia after subtotal gastrectomy for gastric cancer. Aliment Pharmacol Ther. 2013 Sep;38(5):477-89. doi: 10.1111/apt.12402. Epub 2013 Jul 3. PMID 23822578